CLINICAL TRIAL: NCT00870051
Title: Endurant Stent Graft Natural Selection Global Postmarket Registry
Acronym: ENGAGE
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: P#888
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Endurant; Stent Graft; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAA patients: Subjects diagnosed with an AAA who are considered candidates for endovascular repair with Endurant Stent Graft, and who meet the inclusion/exclusion criteria are intended to participate in this registry
  Interventions: Device: Endurant Stent Graft

INTERVENTIONS:
Device: Endurant Stent Graft — Endurant Stent Graft implantation
  Other Names: EVAR

SUMMARY:
The purpose of ENGAGE is to prospectively collect global 'real world' data on the Endurant Stent Graft System from AAA subjects.

DETAILED DESCRIPTION:
The Endurant Stent Graft Natural Selection Global Post-market Registry, ENGAGE is initiated to expand the clinical knowledge base by including 'real world' subjects, applying a minimal amount of subject selection criteria. This subject group may better represent the subject profile treated in actual clinical practice without selecting sub-groups of particular low/high risk or excluding certain diseases. ENGAGE aims at following and documenting the subject selections, diagnostic tools used and treatment interventions chosen by the vascular surgeon or interventional radiologist. ENGAGE will not impose CIP required study procedures affecting clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or minimum age as required by local regulations
* Indication for elective surgical repair of AAA with an endovascular stent graft in accordance with the applicable guidelines on endovascular interventions and the Instructions for Use of the Endurant Stent Graft System
* Signed consent form ("Patient informed consent Form" or "Patient Data Release Authorization Form"). The subject or legal representative has been informed of the nature of the trial and has consented to participate and authorized the collection and release of his medical information
* Intention to electively implant the ENDURANT Stent Graft System
* Ability and willingness to comply with the CIP.

Exclusion Criteria:

* High probability of non-adherence to physician's follow-up requirements
* Current participation in a concurrent trial which may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with an AAA who are considered candidates for endovascular
Sampling Method: Non-Probability Sample
Enrollment: 1266 (Actual)
Dates: Start 2009-04-08 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Treatment Success | 10 years

SECONDARY OUTCOMES:
Stent Graft Migration | 10 years
Stent Graft Patency | 10 years
Stent Graft Endoleaks | 10 years
Secondary procedures to correct Type I and III endoleaks | 10 years
Secondary endovascular procedure | 10 years
Adverse Device Effects | 10 years
Technical Observations | 5 years
Aneurysm-related mortality | 10 years
All-cause mortality | 10 years
MAE | 30 days
Health Related Quality of Life Scores | 12 months
Stent Graft Stenosis | 10 years
  Stent Graft stenosis is considered a reduction in the diameter of the stent graft lumen as compared to the reference. SG stenosis will be assessed by imaging as CT with contrast, Ultrasound, etc.
AAA Diameter Increase | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Riambau, Prof., Study Director — Hospital Clinic of Barcelona; Furuzan Numan, prof, Study Director — Memorial Hospital Istanbul; Robert A. Fitridge, Dr., Study Director — The Queen Elizabeth Hospital, Woodville, South Adelaide, Australia; Yehuda Wolf, Prof., Study Director — Tel Aviv Sourasky Medical Center, Israel; Dittmar Böckler, Prof., Study Director — Universtiy of Heidelberg, Germany; Paul Hayes, Dr., Study Director — Addenbrookes Hospital, Cambridge, Great Britain
Locations (80):
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Clínica La Sagrada Familia, Buenos Aires
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - St Andrew's Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Box Hill Hospital, Melbourne, Victoria
  - Epworth Healthcare - Epworth Eastern, Melbourne, Victoria
  - JMLS Medical Services PTY, trading as Perth Institute of Vascular Research, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Hollywood Private Hospital, Perth, Western Australia
- Krankenhaus Hietzing, Vienna, Austria
- Belgium (4):
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint-Blasius-Campus Dendermonde, Dendermonde
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre, Halifax
  - London Health Sciences Centre - Victoria Hospital, London
  - Glen Royal Victoria Hospital, Montreal
  - CHUQ - Hôpital Saint-François d'Assise, Québec
  - Toronto General Hospital, Toronto
- China (3):
  - Chinese PLA General Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - People's Hospital of Guangdong Province, Guangzhou
- Fundacion Cardioinfantil, Bogotá, Colombia
- IKEM - Institutu Klinicke a Experimentalni Mediciny, Prague, Czechia
- France (3):
  - CHU de Bordeaux - Centre Universitaire Pellegrin, Bordeaux
  - Hôpitaux Universitaires - Hôpital Henri Mondor, Créteil
  - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - St. Franziskus-Hospital Münster GmbH, Münster
  - Städtisches Klinikum Solingen, Solingen
- Greece (2):
  - Euromedica - Kyanous Stavros General Hospital, Thessaloniki
  - Papageorgiou General Hospital, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (3):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Ospedaliera-Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Senese, Siena
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Netherlands (6):
  - Rijnstate - Locatie Arnhem, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Zuyderland Medisch Centrum Heerlen, Heerlen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
  - Sint-Elisabeth Ziekenhuis, Tilburg
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato District Health Board, Hamilton
- Norway (3):
  - Helse Bergen HF - Haukeland Universitetssjukehus, Bergen
  - Oslo Universitetssykehus-Rikshospitalet, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
  - Szpital Bielanski, Warsaw
- Hospital de Santa Maria-Centro Hospitalar Lisboa Norte, EPE, Lisbon, Portugal
- Narodny ustav srdcovych a cievnych chorob, a.s. (NUSCH), Bratislava, Slovakia
- South Africa (3):
  - Life Healthcare - Life Kingsbury Hospital, Cape Town
  - Life Healthcare - Life St Georges Hospital, Port Elizabeth
  - Netcare Unitas Hospital, Pretoria
- South Korea (2):
  - Chonnam National University Hospital, Gwangju
  - Yonsei University health System -Severence Hospital, Seoul
- Spain (5):
  - Hospital Universitari Clínic de Barcelona, Barcelona
  - Complejo Hospitalario Universitario Granada Hospital Campus de la Salud, Granada
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset Örebro, Örebro
  - Södersjukhuset, Stockholm
- Inselspital - Universitätsspital Bern, Bern, Switzerland
- Songklanagarind Hospital, Songkhla, Thailand
- Turkey (Türkiye) (4):
  - Istanbul Universitesi - Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Memorial Sisli Hastanesi, Istanbul
  - Dokuz Eylül University, Izmir
  - Adana Baskent University Hospital, Yüreğir
- United Kingdom (5):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge
  - The Royal Liverpool and NHS Broadgreen University Hospitals - Royal Liverpool University Hospital, Liverpool
  - St George's University Hospitals - NHS Trust, London
  - Wythenshawe Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne
- Institucion Medica Uruguaya, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: No
Only multi center data will be available

REFERENCES:
- [Result] Bockler D, Fitridge R, Wolf Y, Hayes P, Silveira PG, Numan F, Riambau V; ENGAGE Investigators. Rationale and design of the Endurant Stent Graft Natural Selection Global Postmarket Registry (ENGAGE): interim analysis at 30 days of the first 180 patients enrolled. J Cardiovasc Surg (Torino). 2010 Aug;51(4):481-91. PMID 20671632
- [Result] Stokmans RA, Teijink JA, Forbes TL, Bockler D, Peeters PJ, Riambau V, Hayes PD, van Sambeek MR. Early results from the ENGAGE registry: real-world performance of the Endurant Stent Graft for endovascular AAA repair in 1262 patients. Eur J Vasc Endovasc Surg. 2012 Oct;44(4):369-75. doi: 10.1016/j.ejvs.2012.07.005. Epub 2012 Jul 24. PMID 22835762
- [Result] Stokmans RA, Teijink JA, Cuypers PW, Riambau V, van Sambeek MR. No differences in perioperative outcome between symptomatic and asymptomatic AAAs after EVAR: an analysis from the ENGAGE Registry. Eur J Vasc Endovasc Surg. 2012 Jun;43(6):667-73. doi: 10.1016/j.ejvs.2012.02.034. Epub 2012 Mar 21. PMID 22440235
- [Result] Dubois L, Novick TV, Harris JR, Derose G, Forbes TL. Outcomes after endovascular abdominal aortic aneurysm repair are equivalent between genders despite anatomic differences in women. J Vasc Surg. 2013 Feb;57(2):382-389.e1. doi: 10.1016/j.jvs.2012.09.075. Epub 2012 Dec 21. PMID 23266281
- [Result] Pol RA, Zeebregts CJ, van Sterkenburg SM, Reijnen MM; ENGAGE Investigators. Thirty-day outcome and quality of life after endovascular abdominal aortic aneurysm repair in octogenarians based on the Endurant Stent Graft Natural Selection Global Postmarket Registry (ENGAGE). J Vasc Surg. 2012 Jul;56(1):27-35. doi: 10.1016/j.jvs.2011.12.080. Epub 2012 Mar 28. PMID 22459746
- [Result] Tang T, Sadat U, Walsh S, Hayes PD; ENGAGE Investigators. Comparison of the endurant bifurcated endograft vs. aortouni-iliac stent-grafting in patients with abdominal aortic aneurysms: experience from the ENGAGE registry. J Endovasc Ther. 2013 Apr;20(2):172-81. doi: 10.1583/1545-1550-20.2.172. PMID 23581758
- [Result] Pol RA, Zeebregts CJ, van Sterkenburg SM, Ferreira LM, Goktay Y, Reijnen MM; Endurant Stent Graft Natural Selection Global Postmarket Registry (ENGAGE) Investigators. Outcome and quality of life after endovascular abdominal aortic aneurysm repair in octogenarians. J Vasc Surg. 2014 Aug;60(2):308-17. doi: 10.1016/j.jvs.2014.02.009. Epub 2014 Mar 20. PMID 24657065
- [Result] Kiguchi MM, Forbes TL, Teijink JA, Pliagas GA, Ellozy SH, Bockler D, Makaroun MS. Clinical application and early outcomes of the aortouni-iliac configuration for endovascular aneurysm repair. J Vasc Surg. 2014 Dec;60(6):1452-9. doi: 10.1016/j.jvs.2014.08.063. Epub 2014 Oct 3. PMID 25282698
- [Result] Faure EM, Becquemin JP, Cochennec F; ENGAGE collaborators. Predictive factors for limb occlusions after endovascular aneurysm repair. J Vasc Surg. 2015 May;61(5):1138-45.e2. doi: 10.1016/j.jvs.2014.11.084. Epub 2015 Feb 2. PMID 25656594
- [Derived] Dijkstra ML, Zeebregts CJ, Verhagen HJM, Teijink JAW, Power AH, Bockler D, Peeters P, Riambau V, Becquemin JP, Reijnen MMPJ; ENGAGE investigators. Incidence, natural course, and outcome of type II endoleaks in infrarenal endovascular aneurysm repair based on the ENGAGE registry data. J Vasc Surg. 2020 Mar;71(3):780-789. doi: 10.1016/j.jvs.2019.04.486. Epub 2019 Aug 20. PMID 31443976
- [Derived] Dijkstra ML, van Sterkenburg SM, Lardenoye JW, Zeebregts CJ, Reijnen MM; ENGAGE Investigators. One-Year Outcomes of Endovascular Aneurysm Repair in High-Risk Patients Using the Endurant Stent-Graft: Comparison of the ASA Classification and SVS/AAVS Medical Comorbidity Grading System for the Prediction of Mortality and Adverse Events. J Endovasc Ther. 2016 Aug;23(4):574-82. doi: 10.1177/1526602816648455. Epub 2016 May 10. PMID 27170150
- [Derived] Broos PP, Stokmans RA, van Sterkenburg SM, Torsello G, Vermassen F, Cuypers PW, van Sambeek MR, Teijink JA. Performance of the Endurant stent graft in challenging anatomy. J Vasc Surg. 2015 Aug;62(2):312-8. doi: 10.1016/j.jvs.2015.03.024. Epub 2015 May 1. PMID 25937606